CLINICAL TRIAL: NCT05749484
Title: Prediction of the Chronicization of Radiation-induced Acute Intestinal Injury Based on the Expression Level of Immune Factors: a Prospective, Observational and Confirmatory Clinical Study
Brief Title: Prediction of the Chronicization of Radiation-induced Acute Intestinal Injury
Acronym: CRAII
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: EC-075
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Radiation-induced Intestinal Injury
Keywords: Chronicization, radiation-induced acute intestinal injury, Rectal cancer, NCRT, TME
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NCRT+TME: Neoadjuvant chemoradiotherapy (NCRT) and total mesorectal excision (TME) Interventions
  Interventions: Other: NCRT+TME

INTERVENTIONS:
Other: NCRT+TME — The eligible patients who voluntarily sign the consent form will undergo NCRT and TME according to treatment guidelines.

SUMMARY:
Our team has constructed a prediction model based on the expression level of immune factors (PD-L1, PD-1, CTLA4, Siglec15) to predict the chronicization of radiation-induced acute intestinal injury (RAII) and verified the predictive efficacy of the system in retrospective studies. This clinical study intends to further prospectively verify the accuracy of this prediction model in rectal cancer patients. In this study, we plan to enroll 200 patients diagnosed with locally advanced rectal cancer by pathology and MRI, who undergo neoadjuvant chemoradiotherapy (NCRT) and total mesorectal excision (TME) and develop RAII during NCRT or within 1 month. We will follow up the occurrence and progression of radiation-induced intestinal injury within 1 year after TME. Expression levels of immune factors will be detected in pathological tissue after TME and applied to the prediction model to predict the chronicization of RAII. Based on the clinical diagnosis of chronic radiation-induced intestinal injury, the area under curve (AUC), accuracy, precision, specificity, and sensitivity of this prediction model in predicting the chronicization of RAII will be evaluated. The main outcome hypothesis is that the AUC of chronicization of RAII predicted by the prediction model based on the expression level of immune factors is more than 0.8.

DETAILED DESCRIPTION:
Study design and setting The study is a prospective, observational, confirmatory, single-center study in predicting the chronicization of radiation-induced acute intestinal injury based on the expression level of immune factors.

Participants Patients diagnosed with locally advanced rectal cancer, who undergo NCRT and TME at The Sixth Affiliated Hospital, Sun Yat-sen University and develop RAII during NCRT or within 1 month will be assessed for suitability for inclusion.

Inclusion criteria Written informed consent. 18-75 years of age. ECOG score for performance status is 0-2. Locally advanced rectal adenocarcinoma (T3-4/N+M0) with pathological and MRI diagnosis. Patient will undergo NCRT and TME therapies and develop RAII during NCRT or within 1 month.

Exclusion criteria Patients with other active malignant tumors. Patients who have received pelvic radiotherapy or immunotherapy. Pathological tissue cannot be obtained after TME. Patients with toxicity (CTCAE Grade ≥ 2) caused by previous treatment that has not subsided. Pregnant or lactating women.

Interventions The eligible patients who voluntarily sign the consent form will undergo NCRT and TME according to treatment guidelines.

Outcomes The primary outcome is the AUC of chronicization of RAII predicted by the prediction model. The secondary outcomes are accuracy, precision, specificity, and sensitivity of this prediction model in predicting chronicization of RAII.

Recruitment Patients aged 18-75 years who have been diagnosed with locally advanced rectal cancer and consider NCRT+TME therapies and develop RAII during NCRT or within 1 month are eligible for the study. The study physicians will inform the patients about the study in detail. After obtaining informed consent, the patient is recruited to the study. We will follow up the occurrence and progression of radiation-induced intestinal injury within 1 year after TME. Expression levels of immune factors will be detected in pathological tissue after TME and applied to the prediction model to predict the chronicization of RAII.

Participant timeline Recruitment started in March 1, 2023 at The Sixth Affiliated Hospital, Sun Yat-sen University.

Sample size We plan to enroll 200 patients diagnosed with locally advanced rectal cancer by pathology and MRI, who undergo NCRT and TME and develop RAII during NCRT or within 1 month.

Data management, collection and monitoring All protocol-required information collected during the study will be entered by the investigator in the electronic case report forms (CRF). The investigator should complete the CRF as soon as possible after information is collected. An explanation should be given for all missing data. The completed CRF will be reviewed and signed by the investigator. The main investigator will continuously monitor data. Data will be stored in the secured network of Sun Yat-sen University and for security reasons, in an external hard drive which will be used to back up regularly the database.

Statistical methods For statistical analysis of the quantitative variables with normal distribution, the mean, standard deviation (SD), median and interquartile range will be calculated. Group comparisons will be made using t tests or Mann-Whitney U test for continuous variables. Associations between the categorical variables will be tested with the Chi-Square-test or the Fisher exact test, when appropriate. Paired values (before and after therapies) will be compared for each patient using a paired t test or a Wilcoxon test. The data will be analyzed using IBM SPSS Statistics for Windows, version 27.0 (IBM Corporation, Armonk, NY, USA). A significance threshold of p < 0.05 will be adopted for all tests.

Research ethic approval The study adheres to the Declaration of Helsinki on medical research protocols and ethics. The protocol was reviewed and approved by the Human Medical Ethics Committee of the Sixth Affiliated Hospital of Sun Yat-sen University (2023ZSLYEC-075).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent. 18-75 years of age. ECOG score for performance status is 0-2. Locally advanced rectal adenocarcinoma (T3-4/N+M0) with pathological and MRI diagnosis. Patient will undergo NCRT and TME therapies and develop RAII during NCRT or within 1 month.

Exclusion Criteria:

* Patients with other active malignant tumors. Patients who have received pelvic radiotherapy or immunotherapy. Pathological tissue cannot be obtained after TME. Patients with toxicity (CTCAE Grade ≥ 2) caused by previous treatment that has not subsided. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced rectal cancer, who undergo NCRT and TME at The Sixth Affiliated Hospital, Sun Yat-sen University and develop RAII during NCRT or within 1 month will be assessed for suitability for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
AUC | 1 year after TME
  Area Under Curve of the prediction model in predicting chronicization of RAII.

SECONDARY OUTCOMES:
Accuracy, precision, specificity, and sensitivity | 1 year after TME
  Accuracy, precision, specificity, and sensitivity of the prediction model in predicting chronicization of RAII.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Long Wang, Ph.D, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fan J, Lin B, Fan M, Niu T, Gao F, Tan B, Du X. Research progress on the mechanism of radiation enteritis. Front Oncol. 2022 Sep 5;12:888962. doi: 10.3389/fonc.2022.888962. eCollection 2022. PMID 36132154
- [Background] MacNaughton WK. Review article: new insights into the pathogenesis of radiation-induced intestinal dysfunction. Aliment Pharmacol Ther. 2000 May;14(5):523-8. doi: 10.1046/j.1365-2036.2000.00745.x. PMID 10792113
- [Background] Lefevre JH, Amiot A, Joly F, Bretagnol F, Panis Y. Risk of recurrence after surgery for chronic radiation enteritis. Br J Surg. 2011 Dec;98(12):1792-7. doi: 10.1002/bjs.7655. Epub 2011 Sep 16. PMID 21928361
- [Background] Hernandez-Moreno A, Vidal-Casariego A, Calleja-Fernandez A, Kyriakos G, Villar-Taibo R, Urioste-Fondo A, Cano-Rodriguez I, Ballesteros-Pomar MD. CHRONIC ENTERITIS IN PATIENTS UNDERGOING PELVIC RADIOTHERAPY: PREVALENCE, RISK FACTORS AND ASSOCIATED COMPLICATIONS. Nutr Hosp. 2015 Nov 1;32(5):2178-83. doi: 10.3305/nh.2015.32.5.9562. PMID 26545675
- [Background] Anwar M, Ahmad S, Akhtar R, Mahmood A, Mahmood S. Antioxidant Supplementation: A Linchpin in Radiation-Induced Enteritis. Technol Cancer Res Treat. 2017 Dec;16(6):676-691. doi: 10.1177/1533034617707598. Epub 2017 May 22. PMID 28532242